CLINICAL TRIAL: NCT01894139
Title: An Optimized Programming of Healthy Children (APPROACH) - The Most Favourable Dietary Protein:Carbohydrate Ratio During Pregnancy in the Context of New Nordic Diet
Brief Title: An Optimized Programming of Healthy Children (APPROACH)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: The Danish Dairy Research Foundation, Denmark (Other); Nordea-Fonden, Denmark (Unknown); LEGO Charity, Denmark (Unknown); Pharma Nord (Industry); Danish Agriculture and Food Council (Other); Danish Pork Levy Foundation (Unknown); The Novo Nordic Foundation (Other)
Responsible Party: Principal Investigator, Christian Mølgaard, Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EFFECT.C02.2012
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pregnancy; Obesity; Gestational Age and Weight Conditions; Maternal Care for Excessive Fetal Growth; Metabolic Disorders
Keywords: Gestational weight gain; Obese women; Fetal programming; Metabolic disorders; Development of obesity; Development og overweight; Complications during pregnancy and birth
MeSH Terms: conditions — Obesity; Metabolic Diseases; Gestational Weight Gain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High-protein/Low-GI Diet (Experimental): High-protein (25-28 E%), especially marine- and dairy-protein (8-10 E%) and low-GI (GI<55) ad libitum Diet in accordance with the principles of palatability and sustainability of the New Nordic Diet.
  Interventions: Other: High-Protein/Low-GI Diet
- Low-protein/High-GI Diet (Active Comparator): Ad libitum diet based on the Danish National Guidelines (NNR) (protein 10-20 E%; no information on restricting glycaemic load (GI ~ 60)) and in accordance with the principles of palatability and sustainability of the New Nordic Diet.
  Interventions: Other: Low-protein/High-GI Diet

INTERVENTIONS:
Other: High-Protein/Low-GI Diet
  Arms: High-protein/Low-GI Diet
Other: Low-protein/High-GI Diet
  Arms: Low-protein/High-GI Diet

SUMMARY:
The Nutrition Research Unit at Copenhagen University Hospital Herlev will during the fall 2013 initiate a randomized and controlled intervention study engaging 390 obese pregnant women. The overall aim of APPROACH is to investigate how an optimal diet during pregnancy influences the programming of the offspring. The children will after birth be included in a prospective cohort according to maternal randomization and examined six times from delivery until the age of nine years.

DETAILED DESCRIPTION:
Overweight and excessive gestational weight gain (GWG) is associated with increased risk of high birth weight; furthermore there is increased risk of the child developing overweight, diabetes and other metabolic diseases in childhood or adulthood. The effect of reducing gestational weight gain while supplying optimized amount and sources of nutrients is not well investigated. Increased knowledge to the possibility and efficacy of preventing overweight and related diseases is necessary. Modification of protein source and increase in ratio of protein in relation to amount of carbohydrate and reduction of glycaemic index (GI) has in observational studies individually been linked to improved fetal body composition, metabolism and weight control later in life, and less weight gain and weight retention for the mother. The overall aim of APPROACH is to investigate how an optimal diet during pregnancy influences the programming of the offspring. This study will increase the knowledge of the effect of a specific nutrient composition and weight retention during pregnancy on growth and development during the foetal stage and until nine years off age, risk markers later metabolic diseases, especially diabetes and metabolic syndrome. APPROACH will be a dietary intervention investigating differences in responds to a high-protein, especially marine and dairy protein and low-GI diet versus a diet according to the Nordic Nutritional Recommendations. All visits and assessment will be performed by trained staff at Copenhagen University Hospital Herlev. Subjects will be women with expected delivery at Department of Gynaecology and Obstetrics and all examinations of gestational development and foetal growth will take place her; assessment of the children will be performed at the Department of Paediatrics. A total of 390 obese (body mass index (BMI) ≥ 28 kg/m2) pregnant women will be randomized to intervention or control and engage in the program from late first trimester or early second trimester to birth. After birth the children will be included in a prospective cohort according to maternal randomization and examined six times from delivery until the age of nine years. APPROACH will increase the knowledge of the effect of a nutrient composition with high protein for carbohydrate ratio and weight retention during pregnancy on growth and development during the foetal stage and until nine years off age, risk markers later metabolic diseases, especially diabetes and metabolic syndrome. Plasma lipids, markers of metabolic diseases, epigenetics and vitamin D status will be assessed at baseline and several times during pregnancy; and in both intervention and control group these data will increase the knowledge of the effect of supplementing with marine oils and vitamin D in pregnant women. Results from the intervention will be communicated to the general population and published in peer-relieved journals.

ELIGIBILITY:
Inclusion Criteria:

* Birth planed at Copenhagen University Hospital Herlev
* Pre-pregnancy BMI 28-45
* Age 18-42 years
* Speak and understand oral and written Danish
* Singleton pregnancy

Exclusion Criteria:

* Multiple pregnancy
* History of spontaneous abortions or gestational diabetes or preeclampsia or spontaneous preterm birth
* Dairy product intolerant or allergic
* > 10 kg weight change during the past year
* Abuse of alcohol or drugs (>14 units of alcohol per week)
* Critical or chronic disease: diabetes, kidney disease, medically treated heart diseases or arthritis, sarcoidosis, tuberculosis, cancer, liver disease, inflammatory gastrointestinal or lung disease, known active metabolic disease.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 280 (Actual)
Dates: Start 2014-01-04 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Gestational weight gain | Gestational week 14, 15, 17, 21, 25, 28, 36, 39
  Changes in bodyweight, body composition (Magnetic Resonance Imaging) and measurements of body fat by means of skinfold thickness and mid-upper arm circumference.

SECONDARY OUTCOMES:
Growth and development of fetus and child | Gestational week 11+2, 14+0, 28, 32, 36 and month 0, 6, 18, 36 and year 5, 9
  Fetus: Nuchal Translucency Scan (once gw 11+3 - 14+0) and ultrasound scan (gw 28, 32, 36); child: Height in meter, weight in kilograms, body composition (Bioimpedance (month 6,18) and Dual-energy X-ray absorptiometry, DXA (month 0, 36, year 5, 9) , and Magnetic Resonance Imaging (year 9)), skin fold thickness and mid-upper arm circumference, IGF-1.
Fetal programming of obesity and metabolic disorders | Month 0, 6,18, 36 and year 5, 9
  Fasting blood samples (month 0 from umbilical cord), not at 6 months and 18 months; continuous glucose monitoring (year 9) in mmol/L; dietary intake, physical activity, growth and development.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Mølgaard, Professor, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Faculty of Sceience, NEXS, Copenhagen, Frederiksberg, Denmark

REFERENCES:
- [Derived] Larson EA, Magkos F, Zingenberg H, Svare J, Astrup A, Geiker NRW. A high protein low glycemic index diet has no adverse effect on blood pressure in pregnant women with overweight or obesity: a secondary data analysis of a randomized clinical trial. Front Nutr. 2023 Nov 21;10:1289395. doi: 10.3389/fnut.2023.1289395. eCollection 2023. PMID 38075210
- See also: Homepage of Department of Nutrition, Exercise and Sports, University of Copenhagen — https://nexs.ku.dk